CLINICAL TRIAL: NCT04599491
Title: INTELLiVENT-ASV Using Mainstream Versus Sidestream End-Tidal CO2 Monitoring- a Randomized Noninferiority Clinical Trial in Cardiac Surgery Patients
Brief Title: INTELLiVENT-ASV Using Mainstream Versus Sidestream End-Tidal CO2 Monitoring
Acronym: INTELLiSTREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Principal investigator and clinical professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: INTELLiSTREAM
Record Dates: First submitted 2020-10-06; First posted 2020-10-22 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Mechanical Ventilation Complication; Intensive Care Unit; Postoperative Care
Keywords: Mechanical Ventilation; INTELLiVENT-ASV; Quality of Breath; Elective Cardiac Surgery; Postoperative Pulmonary Complications; Lung Protective ventilation; Mainstream Capnography; Sidestream Capnography; Noninferiority trial; Closed Loop Ventilation; Intensive Care Unit; Automated Mechanical ventilation

STUDY DESIGN:
Intervention Model Description: INTELLiSTREAM is a single-center randomized clinical noninferiority trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTELLiVENT-ASV with sidestream capnography (Experimental): Patients randomized into the 'Sidestream capnography'-arm will receive postoperative ventilation on the ICU with INTELLiVENT-ASV with sidestream etCO2 monitoring.
  Interventions: Device: Sidestream capnography using the 'Respironics LoFlo Sidestream CO2 Module'
- INTELLiVENT-ASV with mainstream capnography (Active Comparator): Patients randomized into the 'Mainstream capnography'-arm will receive postoperative ventilation on the ICU with INTELLiVENT-ASV with mainstream etCO2 monitoring.
  Interventions: Device: Mainstream capnography using the 'Respironics Capnostat 5 Mainstream CO2 sensor'

INTERVENTIONS:
Device: Sidestream capnography using the 'Respironics LoFlo Sidestream CO2 Module' — Study patients randomized into the 'Sidestream capnography' arm will receive postoperative ventilation on the ICU with INTELLiVENT-ASV with sidestream etCO2 monitoring using the 'Respironics LoFlo Sidestream CO2 Module'.
  Arms: INTELLiVENT-ASV with sidestream capnography
Device: Mainstream capnography using the 'Respironics Capnostat 5 Mainstream CO2 sensor' — Study patients randomized into the 'Mainstream capnography' arm will receive postoperative ventilation on the ICU with INTELLiVENT-ASV with mainstream etCO2 monitoring using the 'Respironics Capnostat 5 Mainstream CO2 sensor'.
  Arms: INTELLiVENT-ASV with mainstream capnography

SUMMARY:
Background

INTELLiVENT-ASV, an automated closed-loop mode of mechanical ventilation, available on Hamilton ventilators for clinical use, uses mainstream end-tidal CO2 (etCO2) monitoring to adjust minute ventilation. However, sensors for mainstream etCO2 monitoring are expensive and fragile. The less expensive and more robust sensors for sidestream etCO2 monitoring could serve as a good alternative to sensors for mainstream etCO2 monitoring.

Objective of the study

The objective of this randomized noninferiority trial is to determine whether INTELLiVENT- ASV with sidestream capnography is noninferior to INTELLiVENT-ASV with mainstream capnography with regard to the percentage of breaths in a broadly accepted predefined 'optimal' zone of ventilation.

Hypothesis

The investigators hypothesize that INTELLiVENT-ASV with sidestream capnography is noninferior to INTELLiVENT-ASV with mainstream capnography with respect to the percentage of breaths a patient spends within the 'optimal' zone of ventilation.

Study design

INTELLiSTREAM is a randomized noninferiority study.

Study population

The study population consists of consecutive elective cardiac surgery patients who are expected to need at least 2 hours of postoperative ventilation in the ICU of Amsterdam Medical University Centers, location 'AMC'.

Intervention

Shortly after arrival at the ICU, patients will be randomized to receive either ventilation with INTELLiVENT-ASV with mainstream capnography or sidestream capnography.

Primary outcome of the study

The primary study endpoint is the percentage of breaths a patient spends inside the 'optimal' zone of ventilation, as defined before (i.e. tidal volume < 10 ml/kg PBW, maximum airway pressure < 30cm H2O, etCO2 between 30-46 mmHg and pulse oximetry between 93-98%).

Secondary outcomes

The percentage of time spent in other ventilation zones, as defined in the protocol. Time to spontaneous breathing, duration of weaning, loss of etCO2 signal, duration of postoperative ventilation and ventilator parameters as well as results of clinically indicated arterial blood gas analysis.

Nature and extent of burden and risks associated with participation, benefit and group relatedness Hamilton ventilators can use mainstream and sidestream etCO2 sensors. INTELLiVENT-ASV is a safe mode of ventilation, also in patients who receive postoperative ventilation. Furthermore, as all patients are sedated as part of standard care during postoperative ventilation, the burden for the patient is minimal

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective cardiac surgery in the Amsterdam University Medical Centers, location 'AMC'
* Planned admission to the ICU for postoperative ventilation
* Expected to need postoperative ventilation for at least 2 hours

Exclusion Criteria:

* Age under 18 years
* Patients previously included in the current clinical trial
* Patients participation in other interventional clinical trials that could influence ventilator settings and ventilation parameters
* Patients with suspected or confirmed pregnancy
* Moribund patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
The percentage (%) of time spent in the 'optimal' zone of ventilation during the first 3 hours of postoperative ventilation using INTELLiVENT-ASV. | During the first 3 hours, since admission on the intensive care unit (ICU) with the start of INTELLiVENT-ASV ventilation mode.
  A breath is considered to be in the 'optimal zone' when the following criteria are met: tidal volume (VT) ≤8 ml/kg predicted body weight (PBW) and maximum airway pressure (Pmax) ≤ 30 cmH2O and end tidal CO2 (etCO2) = 30-46 mmHg and pulse oximetry saturation (SpO2) = 93-98%.
  The ventilation zones are as defined in earlier studies (ClinicalTrials.gov Identifier: NCT03180203)

SECONDARY OUTCOMES:
The percentage (%) of time spent in the 'optimal', 'acceptable' and 'critical' zones during the first 3 hours of postoperative ventilation using INTELLiVENT-ASV. | During the first 3 hours, since admission on the ICU with the start of the INTELLiVENT-ASV ventilation mode.
  An optimal zone as defined under Primary Outcome Measure
  An acceptable zone = VT = 8-12 ml/kg PBW with an etCO2 = 25-30 or 45-50 mmHg, a Pmax = 31-36 cmH2O and a SpO2 = 85-93% or >98%.
  A critical zone = VT >12 ml/kg PBW or an etCO2 = <25 or ≥51 mmHg, a Pmax ≥36 cmH2O or SpO2 <85%.
Time to spontaneous breathing | Time from start of ventilation at the ICU until five or more consecutive spontaneous breaths, assessed up to 30 days.
  Time to spontaneous breathing is defined as the time from start of ventilation at the ICU until five or more consecutive spontaneous breaths.
Duration of weaning | Time from cessation of sedatives and of a rectal temperature > 35.5ºC to tracheal extubation, assessed up to 30 days.
  Duration of weaning is defined as time from cessation of sedatives and of a rectal temperature > 35.5ºC to tracheal extubation.
Duration of postoperative ventilation | Time from start of ventilation at the ICU until tracheal extubation, assessed up to 30 days.
  Duration of postoperative ventilation, defined as time from start of ventilation at the ICU until tracheal extubation
Proportion of failed extubations | Within 48 hours after extubation.
  Failed extubations are defined as re-intubation within 48 hours after extubation and considering only patients who survived and did not undergo re-sternotomy during this time.
Development of postoperative pulmonary complications | During first 5 postoperative days days.
  Postoperative pulmonary complications is collapsed composite of pneumonia, defined as a patient receiving antibiotics and meets at least one of the following criteria: new or changed sputum, new or changed lung opacities on chest radiography when clinically indicated, tympanic temperature > 38.3C, white blood cell count 12,000/mm^3, pneumothorax, defined as air in he pleural space with no vascular bed surrounding the visceral pleura on chest radiography or severe atelectasis, defined as lung opacification with a shift of the mediastinum, hilum or hemidiaphragm towards the affected area, and compensatory over-inflation in the adjacent non-atelectatic lung on chest radiography.
Length of stay in ICU | From admission to ICU to ICU discharge of the patient, assessed up to 30 days.
Readmission to ICU | From admission to ICU to hospital discharge of the patient, assessed up to 30 days.
Mortality in the ICU | From admission to ICU to ICU discharge of the patient, assessed up to 30 days.
Loss of capnography signal | During the first 3 hours, since admission on the ICU with the start of INTELLiVENT-ASV ventilation mode.
  Loss of etCO2 monitoring requiring a correction by ICU nurses.
Incidence of hypoxemia | Time from start of ventilation at the ICU until tracheal extubation, assessed up to 30 days.
  Hypoxemia is defined as percentage of breath with pulse oximetry saturation <85% but only when SpO2 had a quality index >50%.
Ventilatory parameters: pressures | Time from start of ventilation at the ICU until tracheal extubation, assessed up to 30 days.
  Positive end expiratory pressure (PEEP), maximum airway pressure (Pmax) and plateau pressure (Pplat)
Ventilation parameters: volumes | Time from start of ventilation at the ICU until tracheal extubation, assessed up to 30 days.
  Tidal volume (VT) and minute volume (MV)
Ventilation parameters: respiratory rate | Time from start of ventilation at the ICU until tracheal extubation, assessed up to 30 days.
  Respiratory rate (RR)
Ventilation parameters: oxygenation | Time from start of ventilation at the ICU until tracheal extubation, assessed up to 30 days.
  Fraction inspired oxygen (FiO2) and pulse oximetry (SpO2)
Ventilation parameters: capnography | Time from start of ventilation at the ICU until tracheal extubation, assessed up to 30 days.
  End-tidal CO2 (etCO2)
Clinically indicated arterial blood gas analyses | Time from start of ventilation at the ICU until tracheal extubation, assessed up to 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J. Schultz, Prof. dr., Principal Investigator — Amsterdam University Medical Centers location 'AMC'
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing plan will follow

REFERENCES:
- [Derived] Nijbroek SGLH, Roozeman JP, Ettayeby S, Rosenberg NM, van Meenen DMP, Cherpanath TGV, Lagrand WK, Tepaske R, Klautz RJM, Serpa Neto A, Schultz MJ. Closed-Loop ventilation using sidestream versus mainstream capnography for automated adjustments of minute ventilation-A randomized clinical trial in cardiac surgery patients. PLoS One. 2023 Aug 23;18(8):e0289412. doi: 10.1371/journal.pone.0289412. eCollection 2023. PMID 37611007